CLINICAL TRIAL: NCT04348968
Title: Retrospective and Prospective Post-Market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the Zimmer® Maxera™ Cup (Implants and Instrumentation)
Brief Title: Maxera Large Cups - Canada
Acronym: Maxera Canada
Status: Terminated | Type: Observational
Why Stopped: The notified body does not require data anymore and recruitment did not start. The study was thus terminated after approval from the investigator and the local ethical committee.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-15H
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Degenerative Joint Disease of Hip; Osteoarthritis, Hip; Avascular Necrosis of Hip; Post-Traumatic Osteoarthritis of Hip; Congenital Dysplasia of the Hip; Joint Diseases; Rheumatoid Arthritis of Hip
Keywords: Total hip arthroplasty; Medical device; Performance; Safety; Clinical benefits; Hip prosthesis
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Dislocation, Congenital; Joint Diseases | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient who received a Maxera Cup of large diameter: Patient received a Maxera Cup with an outer diameter of 64 mm or 66 mm between Nov 2011 and Feb 2018.
  Interventions: Device: Total hip arthroplasty

INTERVENTIONS:
Device: Total hip arthroplasty — The THA surgical procedure involves replacing the head of the femur and acetabulum or socket with an artificial prosthesis. This system is composed of a femoral stem that is inserted into the femoral canal, a ball that attaches to the femoral stem, and an acetabular component or shell that replaces the acetabulum.
  In this study, the acetabular component is the Zimmer Maxera Cup, which is a monoblock construct consisting of a pre-assembled shell and liner. The ceramic liner articulates with a ceramic femoral head for a ceramic-on-ceramic large diameter head articulation. The Maxera Cup is intended for single use only and is designed for reconstruction of the hip joint for conditions described in the inclusion and exclusion section of this protocol.
  Other Names: Total hip replacement

SUMMARY:
This study is monocentric, retrospective and prospective, non-controlled, consecutive series Post-Market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the Largest Zimmer® Maxera™ Cup (Implants and Instrumentation)

DETAILED DESCRIPTION:
The Zimmer Maxera Cup is a monoblock construct that consists of a preassembled shell and liner. The ceramic liner articulates with a ceramic femoral head for a ceramic-on-ceramic large diameter head articulation.

The BIOLOX® delta ceramic liner (insert) is preassembled to lock into the tapered shell's cavity and articulate with BIOLOX OPTION ceramic femoral heads, sizes 32, 36, 40, 44, and 48 mm and standard BIOLOX delta ceramic femoral head sizes 32, 36, and 40 mm.

This is a single center post-market clinical evaluation. A consecutive series of 32 patients treated with a Maxera Cup (outer diameter 64 mm or 66 mm) between Nov 2011 and Feb 2018 will be identified and invited to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient received a Maxera Cup with an outer diameter of 64 mm or 66 mm.
* The Zimmer Maxera Cup is indicated for non-cemented use in skeletally mature individuals undergoing primary surgery for rehabilitating hips damaged as a result of non-inflammatory degenerative joint disease (NIDJD) including but not limited to osteoarthritis, avascular necrosis, post-traumatic arthritis, congenital hip dysplasia, and inflammatory joint disease (IJD), e.g. rheumatoid arthritis if bone quality is adequate.

Exclusion Criteria:

* Active, old, or remote infection of the hip.
* Osteoradionecrosis.
* Local bone tumors and/or cysts.
* Patients with poor bone quality, where there is inadequate bone to support the implant(s).
* Neuromuscular compromise, vascular deficiency or other conditions in the affected limb that may lead to inadequate skeletal fixation.
* Allergy to the implanted material.
* Patient's physical conditions that would eliminate or tend to eliminate adequate implant support or prevent the use of an appropriately sized implant, e.g. previous surgery, insufficient quality or quantity of bone resulting from conditions such as cancer or congenital dislocation, metabolic bone disease of the upper femur or pelvis, femoral osteotomy revision, girdle stone revision, osteoporosis, osteomyelitis, neuromuscular compromise or vascular deficiency in the affected limb in sufficient degree to render the procedure unjustifiable (e.g. absence of musculoligamentous supporting structures, joint neuropathy) or other conditions that may lead to inadequate skeletal fixation
* Do not use ceramic femoral heads which are not BIOLOX delta or BIOLOX OPTION with Maxera components.
* Use of this device when a less invasive procedure would be sufficient.
* Skeletal immaturity.
* Any nerve or muscle disease that may have a negative effect on gait or weight bearing
* Loss of abductor musculature in the affected limb.
* Poor skin coverage around the hip joint.
* Rapid disease progression as obvious by joint destruction or bone absorption seen on x-ray.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigator provided a list of 32 patients operated consecutively between Nov 2011 and Feb 2018. These patients received the Maxera Cup of outer diameter 64 or 66 mm. The patients have been operated based on the indications and contraindications listed in the Instructions For Use (IFUs) of the implant.
  The investigator will contact these patients to propose study enrollment until he can ensure 20 consecutive THA procedures. He will get their informed consent and retrospectively collect the preop, surgery, immed postop, and 1 year data
  These 20 patients will be followed-up in the frame of the standard clinicla routine and clinical data will be prospectively collected by the investigator at the 5, 7 and 10-year follow-up visits
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Implant survival based on removal or intended removal of the device and determined using the Kaplan-Meier method | 10 years post-surgery

SECONDARY OUTCOMES:
Pain and functional performance based on the Harris Hip Score | 10 years post-surgery
  The score is given from 0 to 100 with Excellent: 90 - 100, Good: 80 - 89, Fair: 70 - 79, and Poor: < 70
Subject quality-of-life determined by the EQ-5D (EuroQoI) score | 10 years post-surgery
  The lowest score (0) corresponds to "the worst health the patient can imagine", and the highest rate (100) corresponds to "the best health he can imagine".
X-rays evaluated for radiolucencies, osteolysis, hypertrophy, subsidence, heterotopic ossification, etc | 10 years post-surgery
Safety based on eventual complications occurred including dislocations and revisions/removals | 10 years post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vivoda, Study Director — Zimmer Biomet
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada